CLINICAL TRIAL: NCT03000595
Title: A Double-Blind, Randomized, Placebo-Controlled, Safety, Tolerability, and Efficacy Trial of a Botanical Drug Product Containing East Indian Sandalwood Oil (EISO) For The Treatment of Atopic Dermatitis
Brief Title: A Trial of a Botanical Drug Product Containing East Indian Sandalwood Oil (EISO) For Treatment of Atopic Dermatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study location changed
Sponsor: Santalis Pharmaceuticals, Inc. (Industry)
Collaborators: ClinDatrix, Inc. (Industry); Fremantle Dermatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAN007-03
Record Dates: First submitted 2016-12-16; First posted 2016-12-22 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Atopic Dermatitis
Keywords: eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAN007 Cream (Experimental): A cream containing 5% East Indian sandalwood oil (EISO).
  Interventions: Drug: SAN007 Cream
- Placebo (Placebo Comparator): A placebo cream containing the same components as the vehicle for the active intervention arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAN007 Cream — A cream containing 5% East Indian sandalwood oil (EISO).
  Other Names: Active
  Arms: SAN007 Cream
Drug: Placebo — The vehicle cream
  Other Names: SAN007 Placebo Cream
  Arms: Placebo

SUMMARY:
This trial will be a double-blind, randomized, placebo-controlled, safety, tolerability and efficacy trial of SAN007 (5% East Indian sandalwood oil in a cream formulation) treatment regimen when administered daily for up to 28 days to patients from 3 months to 65 years of age, with atopic dermatitis.

DETAILED DESCRIPTION:
Patients will enter the Screening Period once the informed consent/ascent and photographic consent process has been completed. Patients with a total body surface area (BSA) of ≥2% and ≤ 15% atopic dermatitis involvement, in the treatable areas, and who meet all of the inclusion and none of the exclusion criteria will be enrolled.

Once patient eligibility is confirmed and the screening procedures completed, the patient will start the Treatment Period of the study. All enrolled patients will receive either 5% SAN007 cream or placebo cream (randomized in a 2:1 ratio) with the first dose applied at the Day 1 Study Visit. Patients and/or their legally authorized representative will be instructed on how to apply the study medication twice daily for 28 days. Patients will return to the clinic on Study Days 7,14 and 28 for study-related assessments. Patients and/or their LAR will receive a telephone contact from the site, on Study Days 21 and 35.

Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug.

In addition cutaneous tolerability will be evaluated at each visit. Tolerability evaluation will be based on patients reporting discomfort during or immediately following application of SAN007. This will also be recorded as an AE. The study exclusion areas are to be not to be used in this evaluation.

Efficacy will be assessed at each study visit through the completion of the IGA, EASI and BSA calculation.

During the active treatment period, Patients will return to the study site according to the study schedule for interim assessments and recording of concomitant medication and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 3 months of age
2. Have atopic dermatitis, as determined by an EASI score of ≥5 and ≤50 (Hanifin, 2001)
3. Total treatment area(s) of atopic dermatitis involvement ≥2% and ≤10% body surface area (BSA).
4. Have atopic dermatitis that has been clinically stable for ≥ 1 month prior to the Screening Visit.
5. Are able to obtain written informed consent/ascent in a manner approved by the Institutional Review Board and comply with the requirements of the study.
6. Are willing to refrain from using any lotions, moisturizer, cleansers, cosmetics or creams, other than those issued as part of the study, on the target treatment areas during the treatment period.
7. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events.
8. Are willing to refrain from exposure to artificial ultraviolet radiation for the duration of the study.
9. Are willing to cover target treatment areas to avoid exposure to natural ultraviolet radiation for the duration of the study.
10. If female of childbearing potential, must be willing to practice an acceptable form of birth control for the duration of the study. i.e. barrier method, hormone or intrauterine device.
11. Are willing to avoid participation in any other clinical trial for the duration of this study.
12. Are willing to refrain from treating areas that are not the defined treatment area(s), which will be excluded from all assessments and BSA calculation.
13. Are willing to refrain from treating study restricted areas. Study restricted areas are as follows: head, neck, soles of feet, palms of hands, axillae, or intertriginous areas.

Exclusion Criteria:

1. Have a sibling or immediate family member already participating in this trial.
2. Currently requires and/or, in the past month, has required topical use of a medium or high potency steroid.
3. Atopic dermatitis that, in the opinion of the investigator, is likely to stem from an allergic reaction. (i.e. contact dermatitis)
4. Have <2% of atopic dermatitis involvement eligible for treatment.
5. Have participated in any interventional clinical trial in the previous 30 days to the screening visit.
6. Have a known sensitivity to any of the constituents of the test product including sensitivities to sandalwood oil, fragrances or any member of the Compositae family of vascular plants (e.g., sunflowers, daisies, dahlias, etc.).
7. Have received phototherapy within the last 2 months prior to enrollment.
8. Have received any systemic medication for atopic dermatitis in the past 2 months that would interfere with the evaluation of atopic dermatitis (excluding antihistamines or leukotriene inhibitors).
9. Have a present condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
10. Are pregnant, breast-feeding or plan to become pregnant at any point for the duration of the trial.
11. Are not willing to practice an approved form of birth control while on the study drug for the duration of the trial. i.e. barrier method, hormone or intrauterine device.
12. Have been treated, with prescription medication for atopic dermatitis, with no improvement in condition, within 60 days prior to the Baseline visit.
13. Have any evidence of systemic cancer, squamous cell carcinoma, basal cell carcinoma, or any other confounding skin condition.
14. Have undergone treatments with topical atopic dermatitis drug products, other than retinoids or corticosteroids, within 14 days prior to the Baseline Visit, and for therapy containing corticosteroids or retinoids within 28 days prior to Baseline Visit.
15. Have open sores or open lesions in the treatment area(s).
16. Have a history of alcohol or illegal drug/substance abuse, or suspected alcohol or illegal drug/substance abuse in the past two years.
17. Require greater than 2.0 mg/day inhaled or intranasal corticosteroids.
18. Have an active infection of any kind at Baseline
19. Have an occupation that requires ≥50% of time be spent outdoors, where prolonged exposure to ultraviolet radiation is unavoidable.

Ages: 3 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug.
Incidence of Irritation or Rash at the Site of Application of the Study Medication | 28 Days
  The percentage of patients reporting discomfort either during or immediately following the application of SAN007.

SECONDARY OUTCOMES:
Percentage of Patients who Achieve an Improvement in Investigator Global Assessment Score | 28 Days
  The number of patients achieving an Investigator Global Assessment of "clear" or "almost clear" at any time point during therapy
Percentage of Patients who have a ≥ 25% reduction in the Eczema Area and Severity Index (EASI) score | 28 days
  Percentage of patients who have a ≥ 25% reduction in the Eczema Area and Severity Index (EASI) score at any point during the trial.
Percentage of Patients who have a ≥ 50% reduction in the Eczema Area and Severity Index (EASI) score | 28 Days
  Percentage of patients who have a ≥ 50% reduction in the Eczema Area and Severity Index (EASI) score at any point during the trial.
Percentage of patients achieving at least a 1-grade improvement in Investigator Global Assessment score | 28 Days
  Percentage of patients achieving at least a 1-grade improvement in Investigator Global Assessment score
Percentage of patients who have at least a 20% reduction in BSA affected by atopic dermatitis. | 28 Days
  Percentage of patients who have at least a 20% reduction in BSA affected by atopic dermatitis.

IPD SHARING:
Plan to Share IPD: No